CLINICAL TRIAL: NCT06485895
Title: Clinical Evaluation of an IGRA Test for the Diagnosis of Active and Latent Tuberculosis
Acronym: TUBIGRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM24_0100; 2024-A00322-45 (Other: N°IDRCB)
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: TUBERCULOSIS
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TUBERCULOSIS (LATENTE OR ACTIVE) ARM (Experimental)
  Interventions: Diagnostic Test: test IGRA; Diagnostic Test: TEST QUATIFERON TB Gold Plus

INTERVENTIONS:
Diagnostic Test: test IGRA — BLOOD SAMPLES
Diagnostic Test: TEST QUATIFERON TB Gold Plus — BLOOD SAMPLES

SUMMARY:
Methodology This is a single-center study carried out as part of routine patient care.

The aim of the study is to determine the performance of the 2nd generation TB-IGRA test in the diagnosis of tuberculosis.

DETAILED DESCRIPTION:
It is planned to include 500 patients. An enrolment of 455 subjects will enable us to demonstrate sensitivity-specificity levels of 92% for a 95% confidence interval and a 0.05 degree of precision. To take account of non-analyzable samples or tests, the investigator will include 500 subjects

ELIGIBILITY:
Inclusion Criteria:

* Individual at least 18 years of age
* Patient presenting for treatment of tuberculosis disease
* Having undergone or benefiting from screening for tuberculosis using a medically prescribed reference IGRA test.
* Informed patient who has not expressed opposition to participating in the study.

French-speaking patient with unambiguous understanding of oral and written instructions.

Exclusion Criteria:

Persons in a period of exclusion from another study

* Pregnant, parturient or breast-feeding women;
* Person deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity of TB-IGRA 2nd generation test | 24 MONTHS
specificity of TB-IGRA 2nd generation test | 24 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — ASSISTANCE PUBLIQUE HOPITAUX D EMARSEILLE
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No